CLINICAL TRIAL: NCT04172402
Title: A Study of Nivolumab Combination Gemcitabine and S1 as the First-Line Treatment in Patients With Advanced Biliary Tract Cancer
Brief Title: NGS as the First-line Treatment in Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1219
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-09

CONDITIONS: Advanced Biliary Tract Cancer
Keywords: Advanced Biliary Tract Cancer; Nivolumab; Phase 2
MeSH Terms: interventions — titanium silicide; Gemcitabine; Nivolumab

STUDY DESIGN:
Intervention Model Description: Advanced Biliary Tract Cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGS (Experimental): Eligible patients will receive Nivolumab 240mg on day 1, gemcitabine 800 mg/m2/day on day 1 and S-1 orally 80-120 mg/day (depending on patient's body surface area (BSA)) on day 1 to 10 in a 2-week cycle.
  * BSA < 1.25 m2: 80 mg/day
  * 1.25 m2 ≤ BSA < 1.5 m2: 100 mg/day
  * BSA ≥ 1.5 m2: 120 mg/day The treatment will be administered until disease progression, intolerable toxicity, or consent withdrawal during any time of the study.
  Interventions: Drug: TS-1; Drug: Gemcitabine; Drug: Nivolumab

INTERVENTIONS:
Drug: TS-1 — Intervention is administered to patients in this Arm.
Drug: Gemcitabine — Intervention is administered to patients in this Arm.
Drug: Nivolumab — Intervention is administered to patients in this Arm.

SUMMARY:
To evaluate disease objective response rate (ORR) of nivolumab in combination with gemcitabine and TS1 in patients with advanced biliary tract cancer

DETAILED DESCRIPTION:
The primary endpoint will be evaluating overall response rate (ORR) of nivolumab in combination with gemcitabine and TS-1 in patients with advanced BTC. Simon's two-stage design will be used. If there are 3 or fewer subjects with controlled disease in these 19 patients, the study will be stopped. Otherwise, 25 additional patients will be accrued for a total of 44. The null hypothesis will be rejected if 11 or more subjects with controlled disease are observed in 44 patients.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed locally advanced or metastatic biliary tract carcinoma (including intrahepatic bile duct, extrahepatic bile duct, gallbladder and ampulla of vater);
2. no history of chemotherapy or radiotherapy for biliary tract cancer, except those delivered as adjuvant setting that completed at least 6 months before documentation of recurrence by imaging study.
3. presence of at least one measurable tumor lesion which is defined as lesions that can be accurately measured in at least 1 dimension with longest diameter (LD) ≥20 mm using conventional techniques or ≥10 mm with spiral CT and MRI; measurable lymph nodes must be ≥15 mm in the short axis;
4. adequate hematopoietic function which is defined as below:

   1. hemoglobin level ≥ 9 g/dL;
   2. absolute neutrophil count (ANC) ≥ 1,500/mm3;
   3. platelet count ≥ 100,000/mm3;
5. adequate hepatic function which is defined as below:

   1. total bilirubin < 2 mg/dL;
   2. Alanine aminotransferase (ALT) ≤ 3 x ULN; ≤ 5 x ULN if liver metastasis
6. adequate renal function: creatinine clearance rate (CCr) ≥ 50 mL/min ((based upon Cockroft-Gault formula or 24-hour urine collection); < Cockroft-Gault formula > Male: ((140 - age) × weight [kg])/(72 × serum creatinine[mg/dL]) Female: 0.85 x estimate for male
7. age of 20 years or above;
8. ECOG performance status 0-1;
9. life expectancy of at least 12 weeks;
10. patients with childbearing potential shall have effective contraception for both the patient and his or her partner during the study.
11. ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. other malignancy within the past 5 years except for adequately treated basal or squamous cell skin cancer or cervical cancer in situ;
2. history or known presence of brain metastasis;
3. presence of grade 2 or above ascites or pleural effusion;
4. presence of grade 2 or above diarrhea;
5. presence of mental disease or psychotic manifestation;
6. active or uncontrolled infection;
7. significant medical conditions that is contraindicated to study medication or render patient at high risk from treatment complications based on investigator's discretion;
8. pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential.
9. History of active autoimmune disease within 3 years or long-term use of steroid more than prednisolone 10mg/day.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 1 year
  To evaluate disease objective response rate (ORR) of nivolumab in combination with gemcitabine and TS1 in patients with advanced biliary tract cancer

CONTACTS AND LOCATIONS:
Overall Officials: Chen Ming-Huang, MD, Study Chair — Taipei Veterans General Hospital, Taipei, TAIWAN; Chiang Nai-Jung, MD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (6):
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Linkou District
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Chiang NJ, Tang CY, Bai LY, Chang PC, Chen WM, Kang ST, Chen SC, Chen MH, Hsieh JC. Circulating miRNAs as potentially predictive biomarkers for chemoimmunotherapy in advanced biliary tract cancer: a post-hoc analysis of the phase II T1219 study. NPJ Precis Oncol. 2025 Aug 30;9(1):307. doi: 10.1038/s41698-025-01099-x. PMID 40885799